CLINICAL TRIAL: NCT05922007
Title: The Effect of Chronic Pain and Its Treatment on Quality of Life, Disability, and Physical Activity
Brief Title: The Effect of Chronic Pain and Its Treatment on Quality of Life and Physical Activity
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-Chronic Pain; 11/RVO/FNOs/2023 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2023-06-15; First posted 2023-06-28 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pain
Keywords: Pain; Chronic Pain; Health-Related Quality of Life; Physical Activity; Patterns of Activity; Psychological Status; Lower Back Pain
MeSH Terms: conditions — Chronic Pain; Pain; Motor Activity; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Validation study: A total of 150 patients with chronic pain (18-65 years) will be included in the validation of the Czech version of the Patterns of Activity Measures-Pain scale (POAM-P/CZ). The reliability and validity study will have a cross-sectional design.
  Interventions: Other: Validation of the Questionnaire
- Prospective quantitative study: For 150 patients with chronic pain aged 18-65 years, a questionnaire survey will be carried out using the questionnaire set three times, during the first regular check-up at the outpatient clinic and after at least 3 and 6 months, also during a regular check-up.
  Interventions: Other: Prospective quantitative study - questionnaire survey

INTERVENTIONS:
Other: Validation of the Questionnaire — Validation of the Czech version of the Patterns of Activity Measures-Pain scale (POAM-P/CZ)
  Groups: Validation study
Other: Prospective quantitative study - questionnaire survey — A questionnaire survey will be carried out using the questionnaire set three times
  Groups: Prospective quantitative study

SUMMARY:
Chronic pain is pain whose duration usually exceeds a period of three months and standard treatment is ineffective. This pain brings many changes in physical and psychological functioning to the individual and can even lead to a reduction in the quality of life. The main goal of the project is to determine the impact of pain and treatment on the quality of life and patterns of physical activity in patients with chronic pain. Furthermore, evaluate specific changes in quality of life, disability, physical activity, BMI, and body composition after the application of therapeutic and educational measures. Another goal is to validate an assessment tool for assessing the activity patterns of patients with chronic pain. In the first phase, the Czech version of the Patterns of Activity Measures-Pain scale (POAM-P/CZ) will be validated to assess the activity patterns of individuals with chronic pain. Subsequently, a prospective observational study will be carried out with the aim of comparing differences in quality of life, disability, activity patterns, BMI (body composition), and psychosocial variables after the application of targeted treatment measures and educational interventions. The subjective assessment of pain will be supplemented by the assessment of the Analgesia Nociception Index. The results of the project can contribute to the development of effective long-term strategies for the optimization of educational programs to support the self-management of chronic pain and the specific focus of health care.

DETAILED DESCRIPTION:
Chronic pain is defined as pain whose duration usually exceeds a period of three months and standard treatment is ineffective (exceeds the usual time frame of the duration of an acute illness or the expected time of healing of a pathological condition). This pain is harmful and brings many changes to the individual, it can lead to the devastation of the quality of life. One of the dominant secondary effects of chronic pain is a change in the way one performs activities of daily living. The most common changes in activity are avoidance of activities, overexertion, and modulation of the pace of activities. Determining activity patterns is a condition for subsequent targeted educational activities by the nurse. In the Czech Republic, however, there is no specific tool for evaluating movement activities in patients with chronic pain.

The goal of treatment and nursing care for a patient with chronic pain is to reduce pain intensity, achieve appropriate patterns of physical activity and sleep, and improve quality of life. A key step in treatment is the assessment of pain and its impact on functional status and the level of psychosocial relationships.

The main goal of the research is to determine the impact of pain and treatment on the quality of life and physical activity in patients with chronic pain. Other goals include validating the Patterns of Activity Measures-Pain Scale (POAM-P) questionnaire to assess patterns of daily activities of patients with chronic pain in the Czech Republic, to determine the relationship between chronic pain, quality of life, disability in daily activities, physical activity, BMI and mood disorders, compare differences in quality of life, disability, physical activity, BMI and mood disorders after using different therapeutic approaches and education, compare subjective pain assessment and Analgesia Nociception Index (ANI) assessment.

In the first phase of the study, a transcultural validation of the Czech language version of the POAM-P will be carried out according to published recommendations, followed by the creation of a questionnaire set including demographic characteristics, treatment interventions, assessment of the quality of life, disability, mood disorders, and pain intensity in the second phase. Subsequently, 150 patients with chronic pain will be subjected to a questionnaire survey and BMI measurement repeatedly after a minimum of 3 and 6 months during regular outpatient check-ups. The subjective assessment of pain will be supplemented by the assessment of the Analgesia Nociception Index.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pain lasting at least 3 months
* Age 18-65 years
* Diagnosis of back pain, joint pain in arthrosis, postoperative and post-traumatic pain, and pain in rheumatic diseases
* Czech language competency
* Consent to the research investigation

Exclusion Criteria:

* Severe sight or hearing impairment or other illness that does not allow filling in the questionnaires
* Oncological disease

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain treated at the Centre for Treatment of Chronic Pain at the Department of Anaesthesiology, resuscitation and intensive medicine, University Hospital Ostrava will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life - BREF version (WHOQOL-BREF) | 24 months
  Assessment of the World Health Organization Quality of Life - BREF. Assessment of the effect of pain and its treatment after 3 and 6 months of therapeutic and educational activities in 4 domains: physical health, experience, social relationships, environment and two separate items assessing overall quality of life and health satisfaction. A higher score indicates a higher quality of life.
Oswestry Disability Index (ODI2.1a) | 24 months
  Assessment of the Oswestry Disability Index. Assessment of the effect of pain and its treatment after 3 and 6 months of treatment and educational activities on physical disability (restriction of the ability to sit, stand, lift loads and walk), social handicap (social life, sex life - if relevant, travel, personal care), pain and sleep (10 items). The rating for each item is 0-5 points, maximum 50 points. The resulting score is evaluated as minimal disability, moderate disability, severe disability and paralysis.
Patterns of Activity Measures-Pain scale | 24 months
  Assessment of the Patterns of Activity Measures-Pain scale (POAM-P) after 3 and 6 months of treatment and educational activities. Assessment of the effect of pain and its treatment on physical activities (scores in three areas: Avoidance, Overdoing, and Pacing). Scores for each activity range from 0 to 40 for each behaviour pattern. A higher score indicates a more active individual.
Hospital Anxiety and Depression Scale (HADS) | 24 months
  Assessment of the Hospital Anxiety and Depression Scale consists of two subscales. Each subscale has seven items. The HADS-A (anxiety) subscale measures anxiety symptoms and the HADS-D (depression) subscale measures depression symptoms. HADS-T (total) reflects the overall level of distress. Each item has four answer options, with a possible scoring of 0-3. The total number of points in each scale is 0-21 points. A value of 8 is considered as the cut-off point for mild depression/anxiety and a value of 11 for definite depression/anxiety (11 to 14 - moderate; 15 to 21 - high). The total HADS-T score, which ranges from 0 to 42 points, is also evaluated.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire - Short Form (IPAQ - Short Form) | 24 months
  Assessment of the International Physical Activity Questionnaire - Short Form. The International Physical Activity Questionnaire -Short Form measures free-living physical activity levels. The questionnaire is psychometrically tested and used as an instrument to measure physical activity over the previous seven days of participants. It includes 7 questions that distinguish individuals with high, medium and low physical activity.
Patterns of Activity Measures-Pain scale (POAM-P/CZ) | 24 months
  Trans-cultural validation Patterns of Activity Measures-Pain scale - Czech version (POAM-P/CZ). It consists of 30 questions (10 for each activity pattern: Avoidance, Overdoing, and Pacing). Scores for each activity range from 0 to 40 for each behaviour pattern. A higher score indicates a more active individual.
Pain intensity rating (NRS 0-10) | 24 months
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale 0-10, where 0 is no pain and 10 is the worst pain. The NRS can be administered verbally or in a written format as needed for the patient.
Pain map | 24 months
  The pain map provides the most accurate information about where the patient is in pain. It shows the human body from all sides and some of its parts separately. The patient has the task of marking painful areas. The size of the ring should correspond to the real one area of pain. Colored pencils are used for clarification.
Analgesia Nociception Index (ANI) | 24 months
  Analgesia Nociception Index (ANI) is based on ECG data derived from two single-use ANI electrodes applied in V1 and V5 positions to the chest. The ANI is finally computed from a frequency domain-based analysis of the high frequency component of heart rate variability which also incorporates the respiration rate as a potential confounder. It is displayed as a score from 0-100 with low values reflecting low and high values high parasympathetic predominance in autonomic cardiac control.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Polanská, PhDr., MBA, Study Chair — University Hospital Ostrava; Lucie Sikorová, Assoc.Prof.,PhDr.,Ph.D., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Benaim C, Leger B, Vuistiner P, Luthi F. Validation of the French Version of the "Patterns of Activity Measure" in Patients with Chronic Musculoskeletal Pain. Pain Res Manag. 2017;2017:6570394. doi: 10.1155/2017/6570394. Epub 2017 Feb 1. PMID 28255261
- [Background] Cane D, Nielson WR, McCarthy M, Mazmanian D. Pain-related activity patterns: measurement, interrelationships, and associations with psychosocial functioning. Clin J Pain. 2013 May;29(5):435-42. doi: 10.1097/AJP.0b013e31825e452f. PMID 23247000
- [Background] Suygun ET, Celenay ST. Turkish Translation of the Patterns of Activity Measure-Pain in Patients with Chronic Low Back and Neck Pain: Validity and Reliability. Pain Manag Nurs. 2022 Apr;23(2):231-236. doi: 10.1016/j.pmn.2021.01.008. Epub 2021 Feb 23. PMID 33637433
- See also: The International Physical Activity Questionnaire (IPAQ) website — https://sites.google.com/view/ipaq